CLINICAL TRIAL: NCT00536653
Title: Long Term Changes in Bone Mineral Density and Fracture Risk in Patients Receiving Androgen Deprivation Therapy for Advanced Prostate Cancer, With Stratification of Treatment Based on Presenting Values
Brief Title: Changes in Bone Mineral Density and Fracture Risk in Patients Receiving Androgen Deprivation Therapy for Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wirral University Teaching Hospital NHS Trust (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 55/99
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2007-09-28 (Estimated); Status verified 2007-08

CONDITIONS: Osteoporosis
Keywords: prostate cancer; bone density; osteoporosis; androgen antagonists
MeSH Terms: conditions — Osteoporosis; Prostatic Neoplasms | interventions — bicalutamide; Calcium; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Osteporosis Group (Active Comparator): Patients with a presenting T score < -2.5 (osteoporosis), treated with bicalutamide and Ca/VitD
  Interventions: Drug: Bicalutamide and Calcium/ Vitamin D supplementation
- Osteopenia Group (Active Comparator): Patients with a presenting T score between -1.0 and -2,4 (osteopenia), treated with LHRH agonists and Ca/VitD
  Interventions: Drug: LHRH agonists (Goserelin acetate) and Calcium/ Vitamin D supplementation
- Normal Group (Active Comparator): Patients with a presenting T score > -1.0(normal BMD), treated with LHRH agonists
  Interventions: Drug: LHRH agonists (Goserelin acetate)

INTERVENTIONS:
Drug: Bicalutamide and Calcium/ Vitamin D supplementation — Bicalutamide 150mg once daily, Calcium and Vitamin D supplementation once daily
  Arms: Osteporosis Group
Drug: LHRH agonists (Goserelin acetate) and Calcium/ Vitamin D supplementation — 3 monthly depot injection of LHRH agonist (Goserelin acetate 10.8mg) and Calcium/ Vitamin D supplementation daily
  Arms: Osteopenia Group
Drug: LHRH agonists (Goserelin acetate) — 3 monthly depot injection of LHRH agonists (Goserelin acetate 10.8mg)
  Arms: Normal Group

SUMMARY:
The aim of this study is to determine the long term effects of two types of hormonal treatment for advanced prostate cancer (LHRH agonists and the antiandrogen bicalutamide)on the bone mineral density of patients.

DETAILED DESCRIPTION:
Androgen ablation is the mainstay of treatment for advanced prostate cancer. However,luteinizing hormone-releasing (LHRH) agonists are associated with accelerated bone loss, osteoporosis and fractures. An alternative is the non steroidal antiandrogen, bicalutamide, which acts at the androgen receptor and maintains serum testosterone levels. Our aim was to assess the effects of these two treatments on bone mineral density (BMD) of selected groups of patients, based on their BMD at presentation. All patients will undergo peripheral bone densitometry of the forearm, using dual energy X-ray absorptiometry. Osteoporotic patients, at high risk of fractures, will be commenced on bicalutamide. Osteopenic and normal BMD patients will be commenced on LHRH agonists. All osteopenic and osteoporotic patients will be given calcium and vitamin D supplementation.Patients will undergo annual bone densitometry scans, and will be seen in the clinic every 3 months to monitor well-being and PSA levels. Any patient who fails to respond or escapes treatment with hormone monotherapy will be managed according to the clinical situation by either being switched to a combination of LHRH and bicalutamide or additional oestrogen therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients will locally advanced prostate cancer for whom immediate androgen deprivation was indicated

Exclusion Criteria:

* Previous systemic therapy for prostate cancer
* Patients with any illness or medication that would affect bone and mineral metabolism
* Severe hepatic or renal insufficiency

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 618 (Actual)
Dates: Start 1999-10; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Peripheral Forearm bone mineral density | Over 7 years

SECONDARY OUTCOMES:
Fractures of the thoracolumbar spine | Over 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Nigel J Parr, MBBS, FRCS(Urol), MD, Principal Investigator — Wirral University Hospitals NHS Trust
Locations (1):
- Wirral University Hospitals NHS Trust, Upton, Wirral, Merseyside, United Kingdom